CLINICAL TRIAL: NCT00031837
Title: A Prospective Randomized Controlled Multicenter Study of the Effect of Dalteparin on Quality of Life in Unresectable Pancreatic Cancer
Brief Title: Gemcitabine With or Without Dalteparin in Treating Patients With Unresectable or Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, URCC CCOP Research Base, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069232; URCC-U2200; NCI-5012; NCI-CCC-99-45; NCI-P02-0212
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Cancer; Thromboembolism
Keywords: thromboembolism; stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Thromboembolism | interventions — Dalteparin; Gemcitabine

ARMS (1):
- Dalteparin (Experimental): 5,000 anti-Xa units of dalteparin subcutaneously once daily for six months in addition to gemcitabine at 1,000 mg/m2 as a 30-minute infusion weekly for 7 weeks followed by a week of rest for the first cycle and weekly for three weeks followed by a week of rest for each subsequent cycle.
  Interventions: Drug: dalteparin; Drug: gemcitabine hydrochloride; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: dalteparin
Drug: gemcitabine hydrochloride
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Anticoagulants such as dalteparin may help prevent blood clots in patients being treated with gemcitabine for unresectable or metastatic pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of gemcitabine with or without dalteparin in treating patients who have unresectable or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the quality of life of patients with unresectable or metastatic pancreatic cancer treated with gemcitabine with or without dalteparin.
* Compare the survival of patients treated with these regimens.
* Compare the incidence of venous thromboembolic complications in patients treated with these regimens.
* Determine the safety of dalteparin, in terms of bleeding complications, in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (unresectable nonmetastatic vs metastatic). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes once weekly on weeks 1-7 for the first course only. Beginning on week 9, patients receive gemcitabine IV over 30 minutes once weekly for 3 weeks. Treatment then repeats every 4 weeks for up to 6 months in the absence of unacceptable toxicity or disease progression.
* Arm II: Patients receive gemcitabine as in arm I and dalteparin subcutaneously once daily for 6 months in the absence of unacceptable toxicity.

Quality of life is assessed at baseline and every 4 weeks during study therapy.

Patients are followed every 4 weeks.

PROJECTED ACCRUAL: A total of 400 patients (200 per treatment arm) will be accrued for this study within 40 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma or poorly differentiated carcinoma of the pancreas that is considered ineligible for curative resection

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group 0-2

Life expectancy:

* Not specified

Hematopoietic:

* White Blood Cell count greater than 3,500/mm^3
* Platelet count greater than 100,000/mm^3
* No clinically significant bleeding disorder
* No prior heparin-induced thrombocytopenia

Hepatic:

* Bilirubin less than 2.0 mg/dL
* aspartate aminotransferase less than 3 times normal

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* No prior hemorrhagic stroke
* No uncontrolled hypertension (sustained blood pressure greater than 200 mm Hg systolic or 110 mm Hg diastolic)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy
* No gastrointestinal bleeding within the past 30 days
* No contraindications to anticoagulation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for metastatic disease
* Prior adjuvant chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Prior surgical resection allowed
* At least 4 weeks since prior surgery with non-curative intent and recovered
* More than 30 days since prior neurologic or ophthalmologic surgery

Other:

* At least 2 weeks since prior low-molecular-weight heparin
* More than 30 days since prior experimental therapeutic agent
* No concurrent heparin or warfarin for pre-existing condition

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Quality of life as measured by FACT-Hep version 4 every 4 weeks

SECONDARY OUTCOMES:
Survival
Frequency of symptomatic venous thromboembolic complications
Safety as measured by the occurrence of bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: Kishan J. Pandya, MD, Study Chair — University of Rochester
Locations (13):
- United States (13):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - University of Rochester Cancer Center CCOP Research Base, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Northwest, Tacoma, Washington